CLINICAL TRIAL: NCT04588181
Title: Psychological Group Treatment in Adults With Attention Deficit Hyperactivity Disorder: Development of a Short Cognitive -Behavioral Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Josep Antoni Ramos-Quiroga, Head of Psychiatry Department, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AE)249/2016
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT 6 sessions (Experimental)
  Interventions: Behavioral: cognitive behavioral therapy (CBT)
- CBT 12 sessions (Active Comparator)
  Interventions: Behavioral: cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: cognitive behavioral therapy (CBT) — Cognitive behavioral therapy (CBT) is a psycho-social intervention that aims to improve mental health. CBT focuses on challenging and changing unhelpful cognitive distortions (e.g. thoughts, beliefs, and attitudes) and behaviors, improving emotional regulation, and the development of personal coping strategies that target solving current problems.

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder that begins in childhood and can persist throughout adolescence and adulthood. ADHD affects persistently about 5% of children and adolescents and about 2.5% of adults worldwide. The cognitive behavioral therapy (CBT) has proven to be effective in significantly reducing ADHD-symptoms, maintaining the effects during follow-up.

The aim of this study is to develop and validate a psychological treatment program for adult ADHD-patients consisting of six sessions based on Cognitive Behavioural Therapy (CBT) and to study the effectiveness of the developed program in short and long term.

A total of 90 patients will be randomized to two treatment groups (1:1). One group will receive 12 sessions of CBT and the other group six sessions of brief CBT.

It is expected that the short-term effectiveness of a CBT psychological treatment program of six group sessions will be the same as the response to the CBT psychological treatment program of twelve group sessions in adult ADHD-patients with stable drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient with ADHD
* ADHD rating scale>=24
* CGI> 3
* stable pharmacological treatment

Exclusion Criteria:

* IQ<85
* Bipolar Dissorder, Schizophrenia, Psicotic Disorders, Substance Abuse Disorder, Personality Disorders
* Suicidity Ideation
* Serious Organic desease
* Participate in other Psychological Treatment during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Change in the ADHD-Rating Scale (ADHD-RS) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.
  The ADHD-RS is a 18-items scale self-report version for assessing symptoms for ADHD DSM-IV. It consists of a subscale of inattention (IN, 9-items), another of hyperactivity/impulsivity (H / I, 9-items) and the total (TOT, 18-items). The interviewees are asked about the frequency of the symptoms over the past 6 months. Each item is scored from 0 to 3 points, and the highest scores indicates more severe symptomatology of ADHD.
Change in the Clinical Global Impression - Severity (CGI-S) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.

SECONDARY OUTCOMES:
To assess the severity of ADHD symptons | at Baseline
  Assessed by Connors' Adult ADHD Rating Scales Self-report form (CAARS-S:L)
To assess the severity of ADHD symptons | at Baseline
  Assessed by Connors' Adult ADHD Rating Scales Observer form (CAARS-O-L)
To assess the ADHD symptons at childhood | at Baseline
  Assessed by Wender UTAH Rating Scale (WURS). This is a scale used in the diagnosis of attention deficit hyperactivity disorder based on behaviour and feelings experienced during childhood.
  The self-report questionnaire consists of 61-items, 25 of which are highly relevant items for ADHD (thus used in the scale for ADHD) and can help link childhood symptoms with patterns of behaviour in adulthood.
  The scale is however limited by the capacity of the patient to recall memories from childhood.
  Each of the questions in the retrospective scale has 4 answer choices, awarded points from 0 to 4:
  * Not at all or slightly (0 points);
  * Mildly (1 point);
  * Moderately (2 points);
  * Quite a bit (3 points);
  * Very much (4 points).
  The results range between 0 and 100 when the 25-item scale is used and a cut-off at 46 points was provided. This means that patients who score 46 or above are likely to be diagnosed with attention deficit hyperactivity disorder.
To assess the Health status | at Baseline
  Assessed by SF-36. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Change in the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.
  WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) consist of 36 items. The scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed. The lower the score the more disability. The higher the score the less disability
Change in the Functioning Assessment Short Test (FAST) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.
  It comprises 24 items that assess impairment or disability in six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. It is a likert scale. Each item is scored from 0 to 4. The total scored range is from 0 to 96 with a higher score indicating more disability problems.
Change in the Beck Depression Inventory (BDI-II) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.
  the BDI-II also contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Change in the State-Trait Anxiety Inventory (STAI) | In the 6 sessions group: at 6 weeks, at 12 weeks and at 24 weeks.In 12 session group: at 12 weeks, at 24 weeks and at 36 weeks.
  This inventory is made up of 40 questions and they are rated on a 4-point scale. Low scores indicate a mild form of anxiety whereas median scores indicate a moderate form of anxiety and high scores indicate a severe form of anxiety.

IPD SHARING:
Plan to Share IPD: No